CLINICAL TRIAL: NCT03831100
Title: A Single-Site, Parallel-Group, Randomized-Controlled Pilot Trial Comparing BRIGHT With Active Control in Reducing Body Image Disturbance Among Head and Neck Cancer Survivors (BRIGHT 2.0)
Brief Title: Building a Renewed ImaGe After Head & Neck Cancer Treatment (BRIGHT) 2.0
Acronym: BRIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Evan Graboyes, Associate Professor, Department of Otolaryngology- Head and Neck Surgery, Medical University of South Carolina
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00085204; 1R21CA245941-01A1 (NIH)
Record Dates: First submitted 2019-02-04; First posted 2019-02-05 (Actual); Results first posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-07

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible participants will complete baseline questionnaires measuring BID and psychological, social, and emotional wellbeing. Participants will then be randomized to BRIGHT (n=24) or AC (n=24) and undergo weekly, tablet-based BRIGHT or AC for 5 weeks.
  The BRIGHT intervention consists of 5 weekly, 60-minute, tablet-based, one-one telehealth sessions with a licensed therapist. BRIGHT Therapist: A licensed clinical psychologist with extensive experience managing pyscho-oncologic concerns in patients with HNC will deliver BRIGHT.
  The control intervention in this study will be matched to replicate the frequency, intensity, and delivery method of BRIGHT. Participants in the AC arm will thus undergo 5 weekly, 60-minute, tablet-based video sessions in which they undergo non-manualized discussions with a non-trained member of the study team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRIGHT (Experimental): The BRIGHT intervention consists of 5 weekly, 60-minute, tablet-based, one-one telehealth sessions with a licensed therapist. BRIGHT Therapist: A licensed clinical psychologist with extensive experience managing pyscho-oncologic concerns in patients with HNC will deliver BRIGHT.
  Interventions: Behavioral: BRIGHT
- Active Control (Placebo Comparator): The control intervention in this study will be matched to replicate the frequency, intensity, and delivery method of BRIGHT. AC consists of 5 weekly sessions of videos about HNC survivorship that are delivered using a telemedicine platform. Each AC session is a compilation of shorter videos featuring HNC survivors, caregivers, and oncologists discussing non-body image aspects of HNC survivorship.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: BRIGHT — The BRIGHT intervention consists of 5 weekly, 60-minute, tablet-based, one-one telehealth sessions with a licensed therapist. BRIGHT Therapist: A licensed clinical psychologist with extensive experience managing pyscho-oncologic concerns in patients with HNC will deliver BRIGHT.
  Arms: BRIGHT
Behavioral: Active Control — AC consists of 5 weekly sessions of videos about HNC survivorship that are delivered using a telemedicine platform. Each AC session (Table 5) is a compilation of shorter videos featuring HNC survivors, caregivers, and oncologists discussing non-body image aspects of HNC survivorship.
  Arms: Active Control

SUMMARY:
Head and neck cancer (HNC) survivors with body image-related distress (BID) will be randomized to 5-weeks of tablet-based BRIGHT or tablet-based active control (AC; electronic information about HNC recovery). Participants will complete validated measures of BID and psychological, social, and emotional wellbeing to assess the preliminary clinical impact of BRIGHT on BID in HNC survivors. Participants will also complete validated measures of body image coping behavior to assess the role of image coping behavior as the behavioral mechanism of BRIGHT.

DETAILED DESCRIPTION:
Following screening and informed consent, eligible participants will complete baseline questionnaires measuring BID and psychological, social, and emotional wellbeing. Participants (n=44) will then be randomized 1:1 to BRIGHT or AC and undergo weekly, tablet-based BRIGHT or AC for 5 weeks.

The BRIGHT intervention consists of 5 weekly, 60-minute, tablet-based, one-one telehealth sessions with a licensed therapist. The control intervention will be matched to replicate the frequency, intensity, and delivery method of BRIGHT. Participants in the AC arm will thus undergo 5 weekly, 60-minute, tablet-based video sessions in which they undergo non-manualized discussions with a non-trained member of the study team.

Following randomization, patients in each arm will receive a study-issued, cellular-enabled iPad loaded with Vidyo, a video teleconference platform that allows the participant to connect to the study psychologist (BRIGHT) or AC. Vidyo allows face-face communication for tele-cognitive behavioral therapy (CBT) for HNC patients who can articulate well, but also includes a within-video text message feature for aphonic (due to surgical removal of the larynx) or severely dysarthric (due to surgical removal of a significant amount of the tongue) HNC patients who are unable to participate in tele-CBT by speaking. The study iPads are locked to prevent downloading of additional applications. Participants receive a pictorial instructional booklet for logging on to Vidyo. No user names, logins, or web addresses are necessary to connect to the BRIGHT session. The participant simply clicks on the Vidyo application which takes the participant to the assigned teleconference room. At the conclusion of the 5-week intervention, participants return iPads to the study team in pre-addressed, stamped, padded mailers that are provided to the patient.

ELIGIBILITY:
Inclusion Criteria

1. Age > 18 years at the time of screening
2. History of pathologically confirmed invasive squamous cell carcinoma (or histologic variant) of the upper aerodigestive tract (oral cavity, pharynx, larynx, nose/paranasal sinuses), carcinoma of a major or minor salivary gland, or cutaneous malignancy of the face or neck
3. History of curative intent surgery with or without adjuvant therapy, with or without reconstruction
4. American Joint Committee on Cancer (AJCC) 8th Edition pathologic stage grouping I-IV
5. Completion of oncologic treatment within 12 months of study enrollment (but no sooner than 6 weeks post-treatment completion)
6. No planned significant HNC ablative or reconstructive surgery (defined by a postoperative inpatient stay of at least three days) during the study intervention or follow-up period as determined by the HNC oncologic surgeon at the time of study accrual
7. Willingness to be randomized to either BRIGHT or AC
8. Body Image Scale (BIS) score >/= 10

Exclusion Criteria:

1. Inability to speak or write English
2. Pre-existing, ongoing CBT services for other disorders and the participant is not willing to discontinue the prior therapy for the duration of the proposed trial.
3. Initiation or adjustment (< 3 months of baseline) of psychotropic medication.
4. Severe psychiatric comorbidity (e.g. suicidal ideation, psychosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan M Graboyes, MD, MPH, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Graboyes EM, Kistner-Griffin E, Hill EG, Maurer S, Balliet W, Williams AM, Padgett L, Yan F, Rush A, Johnson B, McLeod T, Dahne J, Ruggiero KJ, Sterba KR. Mechanism underlying a brief cognitive behavioral treatment for head and neck cancer survivors with body image distress. Support Care Cancer. 2023 Dec 16;32(1):32. doi: 10.1007/s00520-023-08248-7. PMID 38102496
- [Derived] Graboyes EM, Kistner-Griffin E, Hill EG, Maurer S, Balliet W, Williams AM, Padgett L, Yan F, Rush A, Johnson B, McLeod T, Dahne J, Ruggiero KJ, Sterba KR. Mechanism Underlying a Brief Cognitive Behavioral Treatment for Head and Neck Cancer Survivors with Body Image Distress. Res Sq [Preprint]. 2023 Sep 6:rs.3.rs-3303379. doi: 10.21203/rs.3.rs-3303379/v1. PMID 37720013
- [Derived] Graboyes EM, Kistner-Griffin E, Hill EG, Maurer S, Balliet W, Williams AM, Padgett L, Yan F, Rush A, Johnson B, McLeod T, Dahne J, Ruggiero KJ, Sterba KR. Efficacy of a brief cognitive behavioral therapy for head and neck cancer survivors with body image distress: secondary outcomes from the BRIGHT pilot randomized clinical trial. J Cancer Surviv. 2025 Feb;19(1):140-148. doi: 10.1007/s11764-023-01454-6. Epub 2023 Aug 29. PMID 37644354
- [Derived] Graboyes EM, Kistner-Griffin E, Hill EG, Maurer S, Balliet W, Williams AM, Padgett L, Yan F, Rush A, Johnson B, McLeod T, Dahne J, Ruggiero KJ, Sterba KR. Efficacy of a Brief Cognitive Behavioral Therapy for Head and Neck Cancer Survivors with Body Image Distress: Secondary Outcomes from the BRIGHT Pilot Randomized Clinical Trial. Res Sq [Preprint]. 2023 Aug 7:rs.3.rs-3222601. doi: 10.21203/rs.3.rs-3222601/v1. PMID 37609318
- [Derived] Graboyes EM, Maurer S, Balliet W, Li H, Williams AM, Osazuwa-Peters N, Yan F, Padgett L, Rush A, Ruggiero KJ, Sterba KR. Efficacy of a Brief Tele-Cognitive Behavioral Treatment vs Attention Control for Head and Neck Cancer Survivors With Body Image Distress: A Pilot Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2023 Jan 1;149(1):54-62. doi: 10.1001/jamaoto.2022.3700. PMID 36454561

RESULTS

PARTICIPANT FLOW:
Groups:
- BRIGHT: BRIGHT is video tele-cognitive behavioral therapy delivered one-one for five weekly 60-minute sessions by a licensed clinical psychologist.
- Active Control: Active Control (AC) is a tele-supportive care intervention delivered one-on-one for five weekly sessions via video telemedicine platform.
Period: Overall Study
Arm/Group | BRIGHT | Active Control
Started | 26 | 28
Completed | 20 | 24
Not Completed | 6 | 4
Not completed — Patients who developed a recurrent or new primary cancer went off study per protocol | 6 | 4

BASELINE CHARACTERISTICS:
Population: The efficacy analysis population consisted of all eligible, randomized, evaluable patients. Patients who developed a recurrent or new primary cancer went off study per protocol and were not evaluable.
Groups:
- BRIGHT: The BRIGHT intervention consists of 5 weekly, 60-minute, tablet-based, one-one telehealth sessions with a licensed therapist.
- Active Control: AC consists of 5 weekly sessions of videos about head and neck cancer (HNC) survivorship that are delivered using a telemedicine platform.
- Total: Total of all reporting groups
Arm/Group | BRIGHT | Active Control | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Continuous [Median (Full Range); unit: years] | 63 [31 to 83] | 62.5 [41 to 76] | 63 [31 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 28 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 23 | 22 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 28 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Image Scale Score From Baseline to 1-month Post-intervention
Description: The Body Image Scale (BIS) is a validated, 10-item patient-reported outcome measure (PROM) that assesses the affective, cognitive, and emotional aspects of body image due to cancer or its treatment over the prior 7 days. Responses include 'not at all', 'a little', 'quite a bit', and 'very much', and are scored from 0-3, respectively. Total BIS scores can range from 0-30, with higher scores indicating greater body image dissatisfaction.
Time Frame: 1 month
Population: The efficacy analytic population consisted of all eligible, randomized, evaluable patients. Patients who developed a recurrent or new primary cancer went off study per protocol and were not evaluable.
Measure: Mean (90% Confidence Interval); unit: score on a scale
Groups:
- Active Control: AC is a tele-supportive care intervention delivered one-on-one for five weekly sessions via video telemedicine platform.
Arm/Group | BRIGHT | Active Control
Number analyzed (Participants) | 20 | 24
score on a scale | -3.5 [-5.4 to -1.5] | -0.7 [-2.8 to 1.5]
Statistical Analysis 1: Comparison: BRIGHT vs Active Control; Test type: Superiority; p = 0.25, Regression, Linear — A two-sided P < .10 indicates the a priori threshold for statistical significance. P-values are not adjusted for multiple comparisons; Mean Difference (Net) = -2.1, 90% CI 2-sided [-5.0 to 0.9] — The mean for each study arm represents the mean difference in the score at the post-treatment timepoint relative to the score at baseline. The mean difference (net) represents the mean model-based difference between study arms

2. Secondary Outcome: Change in Body Image Scale Score From Baseline to 3-months Post-intervention
Description: The BIS is a validated, 10-item patient-reported outcome measure that assesses the affective, cognitive, and emotional aspects of body image due to cancer or its treatment over the prior 7 days. Responses include 'not at all', 'a little', 'quite a bit', and 'very much', and are scored from 0-3, respectively. Total BIS scores can range from 0-30, with higher scores indicating greater body image dissatisfaction.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | BRIGHT | Active Control
Number analyzed (Participants) | 20 | 24
score on a scale | -7.3 [-9.7 to -4.8] | -1.6 [-3.9 to 0.7]
Statistical Analysis 1: Comparison: BRIGHT vs Active Control; Test type: Superiority; p = .006, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -5.8, 90% CI 2-sided [-9.1 to -2.5] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change in IMAGE-HN Score From Baseline to 1-month Post-intervention
Description: The IMAGE-HN is a psychometrically sound, 24-item, multi-domain PROM consisting of 4 sub-scales and a global scale that can be used to measure key aspects of HNC-related body image distress (BID) due to HNC or its treatment. Responses include 'Never', 'Rarely', 'Sometimes', 'Often', 'Always', corresponding to a Likert scale of 0-4, respectively. Total IMAGE-HN scores on the global domain (21 questions) range from 0-84, with higher scores indicated greater HNC-related body image dissatisfaction.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | BRIGHT | Active Control
Number analyzed (Participants) | 20 | 24
score on a scale | -8.1 [-13.4 to -2.8] | 0.5 [-5.3 to 6.4]
Statistical Analysis 1: Comparison: BRIGHT vs Active Control; Test type: Superiority; p = .10, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -7.9, 90% CI 2-sided [-15.9 to 0.0] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change in IMAGE-HN Score From Baseline to 3-months Post-intervention
Description: The IMAGE-HN is a psychometrically sound, 24-item, multi-domain PROM consisting of 4 sub-scales and a global scale that can be used to measure key aspects of HNC-related BID due to HNC or its treatment. Responses include 'Never', 'Rarely', 'Sometimes', 'Often', 'Always', corresponding to a Likert scale of 0-4, respectively. Total IMAGE-HN scores on the global domain (21 questions) range from 0-84, with higher scores indicated greater HNC-related body image dissatisfaction.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | BRIGHT | Active Control
Number analyzed (Participants) | 20 | 24
score on a scale | -17.8 [-24.5 to -11.1] | -1.6 [-7.8 to 4.6]
Statistical Analysis 1: Comparison: BRIGHT vs Active Control; Test type: Superiority; p = .002, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -17.1, 90% CI 2-sided [-25.6 to -8.6]

5. Secondary Outcome: Change in Shame and Stigma Scale Score From Baseline to 1-month Post-intervention
Description: The Shame and Stigma Scale is a 20-item, validated, unidimensional PROM that measures four domains (shame with appearance, stigma, regret, and social/speech concerns) in patients with HNC over the prior 7 days. Responses include 'never', 'seldom', 'sometimes', 'often', and 'all the time' and are scored 0-4, respectively. The total score is calculated by summing the individual responses (except for 4 questions which are reverse scored) and thus ranges from 0-80. Higher scores reflect greater shame and stigma from HNC.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: score on a scale
Groups:
- Active Control: AC consists of 5 weekly sessions of videos about HNC survivorship that are delivered using a telemedicine platform.
Arm/Group | BRIGHT | Active Control
Number analyzed (Participants) | 20 | 24
score on a scale | -4.8 [-8.9 to 0.6] | -1.8 [-5.6 to 1.9]
Statistical Analysis 1: Comparison: BRIGHT vs Active Control; Test type: Superiority; p = 0.30, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -3.4, 90% CI 2-sided [-8.8 to 2.0] — Model-based treatment effect estimated using ANCOVA with change score modeled as a function of treatment group (AC, BRIGHT/Therapist A, BRIGHT/Therapist B), with adjustment for baseline scores

6. Secondary Outcome: Change in Shame and Stigma Scale Score From Baseline to 3-months Post-intervention
Description: as for outcome 5
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | BRIGHT | Active Control
Number analyzed (Participants) | 20 | 24
score on a scale | -10.6 [-15.3 to -5.8] | -1.8 [-6.1 to 2.6]
Statistical Analysis 1: Comparison: BRIGHT vs Active Control; Test type: Superiority; p = 0.005, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Median Difference (Net) = -9.7, 90% CI 2-sided [-15.2 to -4.2] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Change in PROMIS SF v1.0-Depression 8a Score From Baseline to 1-month Post-intervention
Description: PROMIS SF v1.0-Depression 8a is a validated, 8-item measure developed by the NIH to assess self-reported negative mood, views of self, and decreased positive affect and engagement. Items are scored using a 5-point Likert scale from 'never' to 'always' (1-5). Higher scores reflect more severe depressive symptoms.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | BRIGHT | Active Control
Number analyzed (Participants) | 20 | 24
score on a scale | -2.7 [-5.1 to 0.2] | 0.5 [-1.7 to 2.8]
Statistical Analysis 1: Comparison: BRIGHT vs Active Control; Test type: Superiority; p = 0.064, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -3.4, 90% CI 2-sided [-6.4 to 0.4] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Change in PROMIS SF v1.0-Depression 8a Score From Baseline to 3-months Post-intervention
Description: as for outcome 7
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | BRIGHT | Active Control
Number analyzed (Participants) | 20 | 24
score on a scale | -3.1 [-6.1 to -0.1] | 0.9 [-1.8 to 3.6]
Statistical Analysis 1: Comparison: BRIGHT vs Active Control; Test type: Superiority; p = 0.046, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -4.3, 90% CI 2-sided [-7.8 to -0.8] — [estimate comment as in outcome 5, analysis 1]

9. Secondary Outcome: Change in PROMIS SF v1.0-Anxiety 8a Score From Baseline to 1-month Post-intervention
Description: The PROMIS SF v1.0-Anxiety 8a is a validated, 8-item measure developed by the NIH to assess self-reported fear, worry, and hyperarousal46. Items are scored using a 5-point Likert scale from 'never' to 'always' (1-5). The total score is calculated by summing the individual responses and thus ranges from 8-40. Higher scores reflect more severe anxiety.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | BRIGHT | Active Control
Number analyzed (Participants) | 20 | 24
score on a scale | -1.6 [-4.3 to 1.1] | -0.3 [-2.8 to 2.2]
Statistical Analysis 1: Comparison: BRIGHT vs Active Control; Test type: Superiority; p = 0.49, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.5, 90% CI 2-sided [-5.2 to 2.1] — [estimate comment as in outcome 5, analysis 1]

10. Secondary Outcome: Change in PROMIS SF v1.0-Anxiety 8a Score From Baseline to 3-months Post-intervention
Description: as for outcome 9
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | BRIGHT | Active Control
Number analyzed (Participants) | 20 | 24
score on a scale | -3.1 [-5.6 to -0.5] | -0.2 [-2.5 to 2.1]
Statistical Analysis 1: Comparison: BRIGHT vs Active Control; Test type: Superiority; p = 0.14, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -3.1, 90% CI 2-sided [-6.5 to 0.3] — [estimate comment as in outcome 5, analysis 1]

11. Secondary Outcome: Change in PROMIS SF v2.0- Satisfaction With Social Roles and Activities 8a Score From Baseline to 1-month Post-intervention
Description: PROMIS SF v2.0-Satisfaction with Social Roles and Activities 8a is a validated, 8-item, measure developed by the NIH to assess self-reported satisfaction with performing one's usual social roles and activities. Items are scored using a 5-point Likert scale from 'not at all' to 'very much' (1-5). The total score is calculated by summing the individual responses and thus ranges from 8-40. Higher scores reflect greater satisfaction with social roles and activities.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | BRIGHT | Active Control
Number analyzed (Participants) | 20 | 24
score on a scale | 3.0 [0.6 to 5.5] | -1.0 [-3.3 to 1.3]
Statistical Analysis 1: Comparison: BRIGHT vs Active Control; Test type: Superiority; p = 0.082, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 3.2, 90% CI 2-sided [0.2 to 6.3] — [estimate comment as in outcome 5, analysis 1]

12. Secondary Outcome: Change in PROMIS SF v2.0- Satisfaction With Social Roles and Activities 8a Score From Baseline to 3-months Post-intervention
Description: as for outcome 11
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | BRIGHT | Active Control
Number analyzed (Participants) | 20 | 24
score on a scale | 6.2 [3.4 to 9.0] | 2.2 [-0.4 to 4.8]
Statistical Analysis 1: Comparison: BRIGHT vs Active Control; Test type: Superiority; p = 0.15, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 2.7, 90% CI 2-sided [-0.4 to 5.7] — [estimate comment as in outcome 5, analysis 1]

13. Secondary Outcome: Change in PROMIS SF v2.0-Social Isolation 8a Score From Baseline to 1-month Post-intervention
Description: PROMIS SF v2.0-Social Isolation 8a is a validated, 8-item, measure developed by the NIH to assess self-reported perceptions of being avoided, excluded or unknown by others. Items are scored using a 5-point Likert scale from 'never' to 'always' (1-5). The total score is calculated by summing the individual responses and thus ranges from 8-40. Higher scores reflect more severe social isolation.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | BRIGHT | Active Control
Number analyzed (Participants) | 20 | 24
score on a scale | -2.9 [-5.3 to -0.4] | -1.3 [-3.4 to 0.9]
Statistical Analysis 1: Comparison: BRIGHT vs Active Control; Test type: Superiority; p = 0.22, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -2.2, 90% CI 2-sided [-5.2 to -0.7] — [estimate comment as in outcome 5, analysis 1]

14. Secondary Outcome: Change in PROMIS SF v2.0-Social Isolation 8a Score From Baseline to 3-months Post-intervention
Description: as for outcome 13
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | BRIGHT | Active Control
Number analyzed (Participants) | 20 | 24
score on a scale | -3.3 [-5.7 to -0.9] | -1.0 [-3.3 to 1.2]
Statistical Analysis 1: Comparison: BRIGHT vs Active Control; Test type: Superiority; p = 0.093, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -2.9, 90% CI 2-sided [-5.8 to -0.1] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: 4 months
Description: Per protocol, only adverse events defined as any undesirable sign, symptom, medical, psychological, social, or emotional reaction that is definitely, probably, or possibly related to the study intervention were collected,
Arm/Group | BRIGHT | Active Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/24
Other Adverse Events (participants affected / at risk) | 0/20 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT03831100/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT03831100/ICF_001.pdf